CLINICAL TRIAL: NCT04308798
Title: Comparison of Surgical Glove Contamination During Total Knee Arthroplasty Procedure
Brief Title: Comparison of Surgical Glove Contamination During Total Knee Arthroplasty Procedure : a Randomized Controlled Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Weerachai Kosuwon, professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HE611285
Record Dates: First submitted 2020-02-25; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Surgical Glove; Total Knee Arthroplasty; Contamination Rate
Keywords: Total knee arthroplasty; Surgical glove; Contamination rate

STUDY DESIGN:
Intervention Model Description: Comparison contamination rate of surgical glove in control group and surgical glove changing group during total knee arthroplasty procedure
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient and outcome assessor will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): No surgical glove changing during total knee arthroplasty procedure
  Interventions: Procedure: Surgical glove changing
- Treatment 1 group (Experimental): Changing surgical glove after draping and before cementation during total knee arthroplasty procedure
  Interventions: Procedure: Surgical glove changing
- Treatment 2 group (Experimental): Changing surgical glove before cementation during total knee arthroplasty procedure
  Interventions: Procedure: Surgical glove changing

INTERVENTIONS:
Procedure: Surgical glove changing — Changing surgical glove after draping and before cementation during total knee arthroplasty

SUMMARY:
Total knee arthroplasty post-op surgical site infection rate about 0.5- 5% Pre-operative , perioperative and post-operative prevention are importance for reduce surgical site infection The prevention of surgical-site infections (SSIs) is an integral component of nosocomial infection control and a major priority in orthopedic surgery.

Surgical wound contamination must be prevented to avoid patient colonisation by microorganisms during surgery.

Surgical glove changing perioperative can reduce contamination and perforation rate Orthopedic surgery had found contamination rate about 20-28 % Joint replacement procedure found contamination rate about 38-67% of all orthopedic surgery 12% of gloves are contaminated after draping and 24% once patient installation is complete.

We hypothesis that changing surgical glove during total knee arthroplasty can reduce contamination rate on surgical glove.

DETAILED DESCRIPTION:
Total knee arthroplasty post-op surgical site infection rate about 0.5- 5% Pre-operative , perioperative and post-operative prevention are importance for reduce surgical site infection The prevention of surgical-site infections (SSIs) is an integral component of nosocomial infection control and a major priority in orthopedic surgery.

Surgical wound contamination must be prevented to avoid patient colonisation by microorganisms during surgery.

Surgical glove changing perioperative can reduce contamination and perforation rate Orthopedic surgery had found contamination rate about 20-28 % Joint replacement procedure found contamination rate about 38-67% of all orthopedic surgery 12% of gloves are contaminated after draping and 24% once patient installation is complete.

Research question : Does changing surgical glove during total knee arthroplasty can reduce contamination rate on surgical glove?

Population : Patient who schedule for primary total knee arthroplasty in Srinagarind hospital

Inclusion criteria :Patient who schedule for primary total knee arthroplasty in Srinagarind hospital

Exclusion criteria :

Patient factor Patient who had previous open knee surgery Patient who have remote infection at period of surgery for total knee arthroplasty Patient who have lower extremity infection same side at total knee arthroplasty prior 48 hrs Surgical glove factor gross perforation Glove changing not include in criteria for study group

Primary outcome :

-Comparison contamination rate of surgical glove in treatment group and control group

Secondary outcome :

-Contamination rate in draping method period and surgical procedure prior to cementation period in total knee arthroplasty

Study design: a randomized controlled trial

Treatment group glove changing after draping and before cementation glove changing before cementation Control group

-no glove change

Pre-operative protocal

* iv. Cefazolin 1 hour prior to incision
* skin preparation by Betadine scrub
* Draping including entire limb from thigh to foot
* pre-operative hand wash by Betadine scrub for at least 2 minutes Perioperative protocal
* Operating room include horizontal laminar flow
* Use Ansell GAMMEX latex powdered surgical glove for all glove include in this study Post-operative protocal
* antibiotic prophylaxis for 24 hours post-op

The five fingertips of each hand were placed on blood agar immediately before each set of gloves were removed Culture plates were subsequently incubated at 37°C for 48 hours. A single microbiologist reported the results of the culture. The number of colonies counted as the number of colony-forming units (CFU) per dish and types of organisms were recorded

identified all bacterial isolates by using Gram stain coagulase oxidase catalase tests. The degree of contamination was divided into three grades

1. no contamination if there was no growth
2. low contamination where between one and five colonies
3. heavily contaminated if there were more than five colonies

ELIGIBILITY:
Inclusion Criteria:

* Patient who schedule for primary total knee arthroplasty

Exclusion Criteria:

* Patient who had previous history of open knee surgery Patient who have remote infection during period of total knee arthroplasty Patient who have infection around lower extremity at the same site of total knee arthroplasty

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
comparison contamination rate on surgical glove | 30 months from randomization
  Contamination rate on surgical glove during total knee arthroplasty

SECONDARY OUTCOMES:
Contamination rate on surgical glove | 30 months from randomization
  Contamination rate on surgical glove during period after draping and before cementation

CONTACTS AND LOCATIONS:
Overall Officials: Navapong Thitiworakarn, Doctor, Principal Investigator — Orthopaedic Department, Faculty of Medicine, Khon Kaen University
Locations (1):
- Orthopaedic Department, Faculty of Medicine, Khon Kaen University, Muang Khonkaen, Changwat Khon Kaen, Thailand